CLINICAL TRIAL: NCT01924377
Title: Characterization and Elimination of Mother Rotors - A Mechanism-targeted Approach for Catheter Ablation of Atrial Fibrillation
Brief Title: Characterization and Elimination of Mother Rotors
Acronym: CENTRA-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed work place
Sponsor: Maria Cecilia Hospital (Other)
Collaborators: Ettore Sansavini Health Science Foundation (Other); Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCH-01
Record Dates: First submitted 2013-08-02; First posted 2013-08-16 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation
Keywords: AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard circumferential pulmonary vein isolation (CPVI) (Other): standard circumferential pulmonary vein isolation by radiofrequenvy ablation
  Interventions: Procedure: standard circumferential pulmonary vein isolation by radiofrequency ablation catheter
- CPVI + Rotor (Experimental): standard circumferential pulmonary vein isolation + rotors' identification and ablation'
  Interventions: Procedure: CPVI + rotors' identification and ablation

INTERVENTIONS:
Procedure: standard circumferential pulmonary vein isolation by radiofrequency ablation catheter — To perform circumferential pulmonary vein isolation left and right circumferential lines will be created with contiguous focal radiofrequency lesions at a distance >5 mm from the pulmonary vein ostia. Two additional ablation lines will be performed in the posterior left atrium (LA), and an ablation line will be placed in the mitral isthmus to prevent postablation LA flutter. Patients with a history of typical atrial flutter will also undergo cavotricuspid isthmus ablation.
  Other Names: Any commercially available Radiofrequency ablation system;; Any commercially available irrigated tip RF ablation catheter (minimum 4 electrodes);
  Arms: standard circumferential pulmonary vein isolation (CPVI)
Procedure: CPVI + rotors' identification and ablation — In CPVI + Rotor arm, two LA sequential maps will be collected before and after CPVI, respectively. During each map creation, rotor electrograms will be identified by the physician. Rotors will be ablated after collecting the second LA sequential map.
  Arms: CPVI + Rotor

SUMMARY:
Recent clinical studies have shown that atrial fibrillation (AF) in humans might be sustained by localized sources called "mother rotors" which exhibit persistent, fast, and well organized activity during AF and play an important role in the generation and maintenance of the fibrillatory activity. In this study, investigators aim to identify the electrophysiological characteristics of mother rotors during atrial fibrillation in patients with paroxysmal and persistent AF and to test whether ablation of such patient-specific substrates might improve the acute and long-term success of conventional catheter ablation therapy.

DETAILED DESCRIPTION:
The present study is designed as a prospective, single-centre, randomized, single-blind, controlled, 2-arm parallel group trial.

The study will consist of:

i) a two-month screening period; ii) randomization and treatment phase; iii) a follow-up phase lasting up to 24 months. Patients with paroxysmal or persistent atrial fibrillation referred to the centre to undergo catheter ablation procedure will be screened. It is expected that approximately 260 patients will be screened in order to have 234 patients fulfilling inclusion criteria at the end of the screening period. The sample will include 154 patients with paroxysmal AF and 80 patients with persistent AF. Paroxysmal and persistent AF will be defined according to current ESC guidelines.

Patients fulfilling selection criteria, will be informed of the study and asked for participation. The study requirements, including required testing, will be discussed with the subject. A signed Informed Consent Form for study participation must be obtained prior to any study-related procedure. Patients will be given a daily diary for recording AF-related signs and symptoms and instructed to bring it back at the inclusion visit.

Eligible patients will be randomised using a web-based randomization system embedded in the electronic CRF (e-CRF).

A randomization schedule, stratified by AF type, using balanced blocks will be established before the start of the trial.

Patients will be randomised to one of the two ablation procedures:

* standard circumferential pulmonary vein isolation (CPVI)
* CPVI followed by rotors' identification and ablation (CPVI + Rotor.

The acute endpoint for AF ablation procedure is electrical isolation of the pulmonary veins and non inducibility of AF by atrial extrastimuli.

Rotors are defined as fast and persistent electrical activation with intracardiac electrograms of regular cycle lengths shorter than 240 ms with stable isoelectric line between two adjacent activation.

The acute endpoints for rotors are their identification by predefined mapping characteristics and their elimination by radiofrequency ablation after circumferential pulmonary vein isolation.

Antiarrhythmic medications may be continued for the first 3 months following the first ablation to avoid early recurrences. At 3 months, antiarrhythmics must be stopped to assess for clinical recurrence.

Freedom from symptomatic AF, atrial tachycardia, and atrial flutter off antiarrhythmic drug therapy as assessed from the end of the 3 months blanking period to 12 months following the ablation procedure, and documented by implantable loop recorder monitoring or trans-telephonic (TT) ECG monitoring.

AF episodes > 10 minutes documented by implantable loop recorder registrations or daily trans-telephonic (TT) ECG will be recorded in the e-CRF, clearly identified by date and time of occurrence. Total duration of the episode will also be recorded. In addition, presence of symptoms, as reported by the patient in the daily diary will be sought.

A Clinical Events Committee (CEC) made up of three cardiologists and arrhythmologists who are not participants in the study will review and adjudicate, symptomatic and asymptomatic AF recurrences.

The Clinical Research Unit staff will support the Investigator and the Sponsor to maintain a high level of ethical, scientific, technical and regulatory quality in all aspects of the Clinical Trial. At regular intervals during the Clinical Trial, the Clinical Research Unit staff will review study progress and any emergent problems. Random source data verification will be performed.

Data will be collected by means of an electronic e-CRF, FDA 21 CFR part 11 compliant.

A detailed Statistical Analysis Plan will be issued.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent atrial fibrillation referred to the centre to undergo catheter ablation procedure
* Age between 18 and 85 years
* Ability to provide informed consent for study participation and be willing and able to comply with study evaluations and follow-up schedule
* AF burden equal to or greater than 24 hours in the screening period before enrollment

Exclusion Criteria:

* Previous AF ablation
* Secondary AF
* Hyperthyroidism
* Left ventricular ejection fraction <30%
* NYHA functional class IV
* Left atrial area > 35 cm2
* Uncorrected severe valvular heart disease
* Contraindication to anticoagulation
* Presence of left atrial thrombus
* Recent (<6 Months) myocardial Infarction or unstable angina or coronary artery by-pass
* Thoracic surgery for congenital, valvular or aortic disease
* History of cerebrovascular accidents
* Pregnancy
* Significant comorbidities such as cancer, severe renal insufficiency requiring hemodialysis, severe obstructive lung disease, cirrhosis, with a life expectancy less than 1 year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05-28 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
freedom from symptomatic AF, atrial tachycardia, and atrial flutter | from the end of the 3 months blanking period to 12 months following the ablation proce
  documented by implantable loop recorder monitoring or trans-telephonic (TT) ECG monitoring

SECONDARY OUTCOMES:
Freedom from asymptomatic AF, atrial tachycardia, and atrial flutter off antiarrhythmic drug | from the end of the 3 months blanking period to 12 months following the ablation procedure
  documented by implantable loop recorder monitoring or trans-telephonic (TT) ECG monitoring
One year clinical/partial success rate | 12 months following the ablation procedure
  defined as a 75% or greater reduction in the number of AF episodes, the duration of AF episodes, or the % time a patient is in AF as assessed with by implantable loop recorder monitoring or trans-telephonic (TT) ECG monitoring measuring AF burden, in the presence or absence of previously ineffective antiarrhythmic drug therapy
Number of Rotors electrograms | at time of pre-ablation electrophysiological mapping
anatomical locations of Rotors electrograms | at time of pre-ablation electrophysiological mapping
characteristics of Rotors electrograms | at time of pre-ablation electrophysiological mapping
  Amplitude and cycle lenght of Rotors electrograms

OTHER OUTCOMES:
a potential relationship between baseline AF burden, number of rotors and outcome | up to 12 months following the ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy